CLINICAL TRIAL: NCT04864210
Title: Analgesia for Video-assisted Thoracoscopic Surgeries: A Comparison Between Intercostal Blocks With Liposomal Bupivacaine and Paravertebral Blocks With Plain Bupivacaine
Brief Title: Video-assisted Thoracoscopic Surgery - Exparel Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nada Sadek (Other)
Collaborators: American Society of Regional Anesthesia (Other)
Responsible Party: Sponsor-Investigator, Nada Sadek, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201901777
Record Dates: First submitted 2021-02-22; First posted 2021-04-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative
Keywords: Video-assisted thoracoscopic surgery (VATS); Paravertebral blocks; Liposomal Bupivacaine (Exparel)
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivacaine (Experimental): The patient will receive an intercostal nerve block by the surgeon in the operating room after anesthetic has been administered. The surgeon will use thoracoscopic guidance to administer the intercostal nerve block. The medication used in this block will liposomal bupivacaine (Exparel).
  Interventions: Drug: Liposomal bupivacaine
- Bupivacaine (Active Comparator): The patient will receive a paravertebral block by the anesthesiologist staffing the pain service area within the hospital prior to surgery. This regional anesthesia will be done using ultrasound guidance. The medication used in this block will be plain bupivacaine with epinephrine.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Surgeons will perform an intercostal nerve block in the operating room under thoracoscopic guidance while the patient is asleep under anesthesia. This intervention (block) is one of the standards of care but the medication (liposomal bupivacaine) currently is not FDA approved for this type of block.
  Arms: Liposomal bupivacaine
Drug: Bupivacaine — An anesthesiologist trained in regional anesthesia will perform a paravertebral block in the hospital's pain service unit. This intervention is standard of care and will use plain bupivacaine with epinephrine as the medication
  Arms: Bupivacaine

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) greatly decreased the number and types of surgery that required open thoracotomy. Initially it was thought that VATS would lead to a reduction of respiratory problems and less acute pain in patients when compared to patients receiving an open thoracic surgery. However, for reasons not clearly understood, a large number of patients who undergo VATS still experience moderate to severe post-surgical pain. Physicians are still faced with the challenge of providing care that will manage both the respiratory issues as well as manage acute pain. The goal of this study is to find the most suitable regimen to effectively manage post-VATS-related pain.

DETAILED DESCRIPTION:
The "promise" was that video-assisted thoracoscopic surgery (VATS) would be associated with less severe pulmonary impairment and less acute post-operative pain compared to open thoracotomy. However, VATS can cause moderate to severe post-operative pain in a significant number of patients and the reason for this is not well understood. In addition it has been found that post-surgical pain can be a strong predictor for the development of chronic pain. Inadequate control of acute pain not only causes serious discomfort and significant respiratory problems, but it may place this population of patients at greater risk of chronic pain and prescription opioid dependence.

Current protocols to manage and/or reduce VATS associated pain include combining the use of regional anesthesia techniques with opioid and non-opioid analgesics. Recent studies have investigated the efficacy of intercostal blocks using liposomal bupivacaine after thoracic surgery. However, these studies lacked an active comparator population of patients.

The study is designed as a prospective randomized study evaluating intercostal blocks using liposomal bupivacaine. The control population of patients will be treated with a paravertebral block using plain bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years and less than 80 years
* Undergoing video-assisted thoracoscopic surgery (VATS) procedure
* BMI less than 40

Exclusion Criteria:

* Unable to provide informed consent
* Non-English speaking
* Pregnant
* BMI greater than 40
* Video-assisted thoracoscopic surgery pleurodesis subjects
* Patients with pre-existing chronic pain
* Opioid tolerance
* Pain syndromes including fibromyalgia, regional pain syndrome or post therapeutic neuralgia in a thoracic distribution
* Allergy to the study medication
* Patients with infectious disease
* Patients with impaired coagulation
* Severe hepatic disease
* Incarcerated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Measure post-operative opioid usage | Up to 48 hours post procedure
  Review the subjects medical record to determine the type and amount of opioid medication that has been taken by the subject in the first 48 hours after surgery,

SECONDARY OUTCOMES:
Measure lung function | Up to 48 hours post procedure
  Using an incentive spirometer device, the amount of air volume inhaled and exhaled by the lungs post VATS procedure. The subject will be asked to do 3 attempts in succession and the number recorded will be the average of the 3 attempts. The air volume inhaled is measured on a scale from near 0 to 2500 milliliters with the low number indicating little air movement whereas 2500 milliliters indicates good air flow. These results will be compared to the volume determined at baseline prior to surgery.
Measure post-operative opioid consumption following discharge from the hospital | Up to 6 months post procedure.
  Patients will be asked to keep a pain medication diary to record their use of opioid and non-opioid medications for pain control.
Measure post-operative pain scores after discharge from the hospital | Up to 6 months post procedure.
  Using a numerical rating scale, patients will be asked to report their pain level. The scale is from 0 to 10 with 0 being no pain and 10 representing the most intense pain. The goal for measuring after acute hospitalization is to determine if the patient is experiencing the onset of chronic pain.
Calculate length of hospital stay | Up to 7 days
  Record the number of days the patients in both arms are hospitalized post VATS procedure. Compare these values between the two groups.
Record the return to normal bowel function | Up to 7 days
  The patient will be asked to report when normal bowel function has returned. It will provide clinicians information as to when other body functions have returned following surgery.
Measure post-operative acute pain scores | Up to 48 hours post procedure
  Using a numerical rating scale (0-10), patients will be asked to report their pain level. The scale is from 0 to 10 with 0 being no pain and 10 representing the most intense pain.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Sadek, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data (IPD) collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.

REFERENCES:
- [Background] Bayman EO, Parekh KR, Keech J, Larson N, Vander Weg M, Brennan TJ. Preoperative Patient Expectations of Postoperative Pain Are Associated with Moderate to Severe Acute Pain After VATS. Pain Med. 2019 Mar 1;20(3):543-554. doi: 10.1093/pm/pny096. PMID 29878248
- [Background] Bayman EO, Parekh KR, Keech J, Selte A, Brennan TJ. A Prospective Study of Chronic Pain after Thoracic Surgery. Anesthesiology. 2017 May;126(5):938-951. doi: 10.1097/ALN.0000000000001576. PMID 28248713
- [Background] Furrer M, Rechsteiner R, Eigenmann V, Signer C, Althaus U, Ris HB. Thoracotomy and thoracoscopy: postoperative pulmonary function, pain and chest wall complaints. Eur J Cardiothorac Surg. 1997 Jul;12(1):82-7. doi: 10.1016/s1010-7940(97)00105-x. PMID 9262085
- [Background] Steegers MA, Snik DM, Verhagen AF, van der Drift MA, Wilder-Smith OH. Only half of the chronic pain after thoracic surgery shows a neuropathic component. J Pain. 2008 Oct;9(10):955-61. doi: 10.1016/j.jpain.2008.05.009. Epub 2008 Jul 16. PMID 18632308
- [Background] Steinthorsdottir KJ, Wildgaard L, Hansen HJ, Petersen RH, Wildgaard K. Regional analgesia for video-assisted thoracic surgery: a systematic review. Eur J Cardiothorac Surg. 2014 Jun;45(6):959-66. doi: 10.1093/ejcts/ezt525. Epub 2013 Nov 27. PMID 24288340
- [Background] Adhikary SD, Pruett A, Forero M, Thiruvenkatarajan V. Erector spinae plane block as an alternative to epidural analgesia for post-operative analgesia following video-assisted thoracoscopic surgery: A case study and a literature review on the spread of local anaesthetic in the erector spinae plane. Indian J Anaesth. 2018 Jan;62(1):75-78. doi: 10.4103/ija.IJA_693_17. PMID 29416155
- [Background] Shariat A, Bhatt H. Successful Use of Serratus Plane Block as Primary Anesthetic for Video-Assisted Thoracoscopic Surgery (VATS)-Assisted Pleural Effusion Drainage. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):e31-e32. doi: 10.1053/j.jvca.2017.10.038. Epub 2017 Oct 31. No abstract available. PMID 29199049
- [Background] Khalil KG, Boutrous ML, Irani AD, Miller CC 3rd, Pawelek TR, Estrera AL, Safi HJ. Operative Intercostal Nerve Blocks With Long-Acting Bupivacaine Liposome for Pain Control After Thoracotomy. Ann Thorac Surg. 2015 Dec;100(6):2013-8. doi: 10.1016/j.athoracsur.2015.08.017. Epub 2015 Oct 24. PMID 26507422
- [Background] Parascandola SA, Ibanez J, Keir G, Anderson J, Plankey M, Flynn D, Cody C, De Marchi L, Margolis M, Blair Marshall M. Liposomal bupivacaine versus bupivacaine/epinephrine after video-assisted thoracoscopic wedge resectiondagger. Interact Cardiovasc Thorac Surg. 2017 Jun 1;24(6):925-930. doi: 10.1093/icvts/ivx044. PMID 28329326
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739